Early initiated vasopressor therapy vs. standard care of primarily fluid therapy in hypotensive patients in the emergency department – A pragmatic, multi-center, superiority, randomized controlled trial Acronym: VASOSHOCK

Statistical Analysis Protocol (SAP) Version 1.0 (15.06.2025)

EU CT identification: 2023-504584-16-00 Clinicaltrials.gov identification: NCT05931601

## **Coordinating Investigator**

Lasse Paludan Bentsen, M.D. Registrar and PhD-fellow in Emergency Medicine

## Sponsor-Investigator

Mikkel Brabrand, M.D., PhD Clinical Professor and Senior Consultant in Emergency Medicine

Research Unit for Emergency Medicine Department of Emergency Medicine Odense University Hospital Kløvervænget 25c, DK-5000 Odense C, Denmark

## Responsible Statistician

Sören Möller, MSc, PhD Professor in Biostatistics Epidemiology, Biostatistics and Biodemography; Department of Public Health, University of Southern Denmark, Odense, Denmark

## Section 1: Administrative Information

This SAP follows the structure suggested by Gamble et al.<sup>1</sup>

## Title and trial registration

1a Descriptive title that matches the protocol, with SAP either as a forerunner or subtitle, and trial acronym (if applicable):

Early initiated vasopressor therapy vs. standard care of primarily fluid therapy in hypotensive patients in the emergency department – A pragmatic, multi-center, superiority, randomized controlled trial

Acronym: VASOSHOCK

Statistical Analysis Protocol (SAP)

## 1b Trial registration number:

EU CT identification: 2023-504584-16-00 Clinicaltrials.gov identification: NCT05931601

#### SAP version

2 SAP version number with dates

Version 1.0 (15.06.2025)

#### Protocol version

3 Reference to version of protocol being used

TRIAL PROTOCOL

Version 2.1

09-12-2025

#### SAP revisions

4a SAP revision history

No revisions yet

4b Justification for each SAP revision

NA

4c Timing of SAP revisions in relation to interim analyses, etc

NA

## Roles and responsibility

## 5 Names, affiliations, and roles of SAP contributors

Coordinating Investigator Lasse Paludan Bentsen, M.D. Registrar and PhD-fellow in Emergency Medicine

Sponsor-Investigator Mikkel Brabrand, M.D., PhD Clinical Professor and Senior Consultant in Emergency Medicine

Research Unit for Emergency Medicine Department of Emergency Medicine Odense University Hospital Kløvervænget 25c, DK-5000 Odense C, Denmark

Responsible Statistician
Sören Möller, MSc, PhD
Professor in Biostatistics
Epidemiology, Biostatistics and Biodemography; Department of Public Health,
University of Southern Denmark, Odense, Denmark

## Signatures of:

Date

Signature

## 6a Person writing the SAP

| Lasse Paludan Bentsen, M.D.<br>Coordinating Investigator | Sören Möller, MSc, PhD<br>Senior statistician | |
|---|---|---|
| Date Signature | Date | Signature |
| 6b Senior statistician responsible | | |
| Sören Möller, MSc, PhD<br>Senior statistician | | |
| Date Signature | | |
| 6c Chief investigator/clinical lead | | |
| Mikkel Brabrand, M.D., PhD<br>Sponsor-Investigator | | |

# Section 2: Introduction Background and rationale

#### From the trial protocol:

Shock is a common occurrence in Danish Emergency Departments (ED)<sup>2</sup> and decreases tissue perfusion while inducing cellular damage and metabolic changes, possibly leading to death<sup>3</sup>. Hypotension, a key component of shock, in the ED is associated with in-hospital mortality of 12% and even higher (33-52%) if identified in the pre-hospital setting.<sup>4</sup> Fluid resuscitation is the most widespread general use for resuscitation of patients with shock,<sup>5,6</sup> but can vary substantially in patients treated in Danish ED's.<sup>7</sup> This is problematic, as liberal fluid resuscitation, such as more than 5 litres over a short period of time, may cause harm<sup>8-11</sup>. When fluid therapy fails, the next step is the initiation of vasopressors such as noradrenaline<sup>12-22</sup>. Noradrenaline applies a primary action on  $\alpha$ -receptors in the blood vessels and partly  $\beta$ -receptors in the heart muscle increasing blood pressure and organ perfusion.<sup>23</sup>

Initiation of peripheral noradrenaline has previously been thought harmful, but newer trials show high safety if handled correctly, while also showing positive outcomes for patients when started early. <sup>13,14,16-22,24-29</sup> In contrast, a delayed vasopressor initiation is associated with increased mortality, even after the first hour of resuscitation. <sup>20</sup> The peripheral administration of noradrenaline provides a shorter time to first infusion, with no increased mortality risk, while still showing a miniscule risk of adverse effects. <sup>12,13,18,21,22,29-31</sup>.

This study will provide evidence if early initiated vasopressor therapy can decrease to time for achieving shock control and subsequentially improve outcomes, such as avoiding ICU admission or reduce length of stay, for some of the most critically ill patients in the Danish ED setting.

#### Aim:

The aim is to investigate whether the use of early initiated vasopressor therapy (i.e., noradrenaline) compared to fluid therapy alone in non-bleeding hypotensive patients presenting in the ED can improve time to shock control and by that, reduce the need for ICU admittance.

## Section 3: Study Methods

## Trial design

This study will be a pragmatic,<sup>32,33</sup> multi-center, superiority, randomized controlled trial, randomizing patients 1:1 to either the intervention group (early vasopressors in the ED) or control group (standard care in the ED).

Adult hypotensive patients who received at least 500ml crystalloid prior to screening will be assessed for eligibility.

The intervention group will receive peripheral infusion of noradrenaline with a starting dose of 0.05 mcg/kg/min and titrated up to a maximum dose of 0.15 mcg/kg/min for up to 24 hours after inclusion.

The standard care group will receive standard care according to local guidelines.

All other treatment considerations are handled at the discretion of the clinical team.

#### Randomization

Patients are randomized in a 1:1 ratio using block randomization by random size of 2, 4, 6 or 8, stratified by trial site. Randomization will be conducted using the web-based randomization system provided in REDCap to ensure allocation concealment.<sup>34</sup>

## Sample size

Described in the protocol.

#### Framework

The trial is a superiority trial.

## Statistical interim analyses and stopping guidance

13a Information on interim analyses specifying what interim analyses will be carried out and listing of time points

No interim analyses are planned

## 13b Any planned adjustment of the significance level due to interim analysis

No interim analyses are planned

#### 13c Details of guidelines for stopping the trial early

No interim analyses are planned

## Timing of final analysis

All analysis will be conducted for all participants when the 30-day follow-up is completed. For the long-term follow-up, this will be conducted after all participants have been assessed for 1-year follow-up and data for this is collected for patients not lost to follow-up.

## Timing of outcome assessments

All data handled during the intervention period is collected at bedside by the clinical staff.

Follow-up data is collected after at least 72-hours and 30-days for the patients.

Consent for participation is collected from the participants, next of kin (of applicable) and the legal guardian as soon as possible after inclusion. In addition, the EQ-5D-5L interview is also collected at this point.

The long-term follow-up data is collected as close as possible to, and at least, 1 year after inclusion.

Outcome assessment times are presented in Table 1:

Table 1: Data collection time points during the trial

| | Screening | Baseline | 24-hours | 72-hours | 30-days |
|-------------------|-------------|----------|----------|----------|---------|
| Time period | Day -2 to 0 | - | 1 | 3 | 30 |
| Consent | | Х | Х | X | Х |
| Randomisation | X | | | | |
| Fluid therapy | Х | | Х | | |
| Vital parameters | X | X | Х | | |
| Vasopressor | | | х | | Х |
| therapy | | | ^ | | ^ |
| SOFA-score at ED | | Х | | (V) | |
| arrival | | ^ | | (X) | |
| Acid-base values | | | | X | |
| ED LOS | | | | Х | |
| AE/SAE | | | Х | Х | |
| Acute Kidney | | х | х | Х | |
| Injury | | ^ | ^ | ^ | |
| Pulmonary | | х | Х | Х | |
| Oedema | | ^ | ^ | ^ | |
| Infection sources | | Х | Х | Х | Х |
| ICU admission | | | | | Х |
| and LOS | | | | | ^ |
| Hospital LOS | | | | | Х |
| Dialysis | | | | | X |
| Non-invasive | | | | | X |
| ventilation | | | | | ^ |
| Invasive | | | | | Х |
| ventilation | | | | | ^ |
| Mortality | | | | | X |
| Readmission | | | | | X |

## Section 4: Statistical Principles

#### Confidence intervals and P values

#### 16 Level of statistical significance

We consider a p-value of < 0.05 statistically significant.

## 17 Description and rationale for any adjustment for multiplicity and, if so, detailing how the type 1 error is to be controlled

We will not perform any adjustment for multiplicity

## 18 Confidence intervals to be reported

We will report 95%CI for all outcomes as specified in section 6.

#### Adherence and protocol deviations

**19a Definition of adherence to the intervention and how this is assessed including extent of exposure** Adherence to the intervention is only considered in the intervention group. Received noradrenaline from the trial during the ED admittance, or department also participating in the trial, will be considered fulfilment of the intervention. The extent of exposure is initiation of noradrenaline at any duration.

The control group receives standard care, and the trial imposes no intervention in this group.

#### 19b Description of how adherence to the intervention will be presented

Exploratory outcomes include any vasopressor treatment at any point within 24 hours, where initiation of the intervention in the intervention group will be presented in this outcome.

The adherence will also be presented in the CONSORT diagram (See Appendix 1: CONSORT diagram draft).

#### 19c Definition of protocol deviations for the trial

Protocol deviations are any deviation of the described trial design in the trial protocol, section 3. This can include: Using other infusion routes than mandated by the trial, not adhering to patient monitoring requirements, treating with noradrenaline past 24-hours post-inclusion and so on.

## 19d Description of which protocol deviations will be summarized

Protocol deviations will be presented with description of number of protocol deviations were reported, including specification of number of patients receiving noradrenaline past 24-hours or at higher doses than allowed.

#### Analysis populations

20 Definition of analysis populations, eg, intention to treat, per protocol, complete case, safety

The trial is analyzed as an intention-to-treat approach for all outcomes in the main analysis. Additional analysis, including safety outcomes are described in

Section 6: Analysis.

## Section 5: Trial Population

## Screening data

All screening data will be presented in text and a trial CONSORT flow-chart. A draft flow-chart can be seen in the appendix.

## Eligibility

#### Inclusion criteria:

- 1. At least 18 years of age
- 2. Signs or suspicion of hypotension or shock (of any type such as septic, vasodilatory or hypovolemic not included in the exclusion criteria) defined as:
  - a. SBP < 100mmHg or MAP < 65 mmHg combined with lactate > 2.0 mmol/L,
  - b. Physician defined blood pressure for the individual patient combined with a lactate > 2.0 mmol/L
  - c. Either SBP < 100mmHg or MAP < 65mmHg with obvious signs of shock with any lactate level evaluated by either two non-specialist physicians (e.g. registrar medical doctors) or one specialist physician.
- 3. Received at least 500ml of intravenous fluid before study inclusion (Including prehospital administration)
- 4. Clinical Frailty Score (CFS) of  $\leq$ 4. If CFS is  $\geq$ 5 and the treating physician find the patient suitable for ICU admittance, the participant can be enrolled, if the on-call ICU doctor would accept the patient for ICU admittance. If the treating physician is unsure of ICU eligibility, regardless of CFS score, the patient should be consulted with the ICU consultant before study inclusion.

#### **Exclusion criteria:**

- 1. Cardiogenic, anaphylactic, haemorrhagic, or neurogenic shock suspected by the treating physician.
- 2. Fertile women (<60 years of age) with positive urine human gonadotropin (hCG) or plasmahCG or women breastfeeding
- 3. Patient deemed terminally ill or with a severe co-morbid status resulting in non-eligibility for ICU admittance decided by either the treating physician or ICU consultant.
- 4. Severe organ failure outside circulatory failure that requires immediate ICU admission.
- 5. Known allergy to noradrenaline.

## 6. Previously enrolled in the trial

#### Recruitment

For a draft CONSORT diagram see appendix 1.

## Withdrawal/follow-up

Participants in the trial can have the intervention terminated before full conclusion of the treatment period. This can include fully termination of participation in the clinical trial including data collection and usage as defined in section 9 and 10.4.4 in the trial protocol. This is considered in the following situations:

- 1. The patient or their legally designated representative withdraws their consent to participate prior to completing the necessary intervention.
- 2. The patients next of kin, for countries where consent can be partly obtained from these, withdraws the consent for the patient to participate prior to completing the necessary intervention. This is only possible, if the patient are yet to provide consent for participation.
- 3. The investigator for safety reasons finds it of best interest of the patient.

In case of early termination of the trial participation and therefore treatment, the clinical staff and investigators must take appropriate steps to ensure the patients treatment and stability of their disease process during early weaning of noradrenaline. This can include quick transfer to the ICU for further treatment of their condition.

Early termination of treatment should be clearly noted, including reason for early termination, in the paper CRF for the patient.

Patients already included, and having consented, to trial participation are expected to complete follow-up, unless they die within the follow-up period.

#### Baseline patient characteristics

Baseline characteristics will be descriptively summarized as proportions (%), mean (SD), median (IQR). Baseline characteristics will not be statistically compared between randomization groups as recommended by CONSORT.<sup>35</sup>

#### The following baseline characteristics will be summarized:

Baseline characteristics will be presented descriptively. No statistical comparisons are carried out for these variables. Expected baseline characteristics are presented in Table 2:

Table 2: Draft of table for baseline characteristics

| Characteristic | | Randomization | |
|---|---|---|---|
| | Overall N = | Early ED vasopressor N = | Standard Care N = |
| Sex | | | |
| Age, years | | | |
| Height, cm | | | |
| Weight, kg | | | |
| Body Mass Index, kg/m2 | | | |
| SBP at ED arrival, mmHg | | | |
| DBP at ED arrival, mmHg | | | |
| MAP at ED arrival, mmHg | | | |
| Pulse at ED arrival, /min | | | |
| SI at ED arrival | | | |
| <0.7 | | | |
| 0.7-0.9 | | | |
| >1 | | | |
| Respiratory rate at ED arrival, /min | | | |
| Oxygen saturation at ED arrival, % | | | |
| GCS at ED arrival | | | |
| Temperature at ED arrival, Celcius | | | |
| SOFA-score at ED arrival | | | |
| Fluid therapy before inclusion, mL | | | |
| Lactate at inclusion, mmol/L | | | |
| <2 | | | |
| ≥2 to <4 | | | |
| ≥4 | | | |
| SBP at inclusion, mmHg | | | |
| DBP at inclusion, mmHg | | | |
| MAP at inclusion, mmHg | | | |
| Infection | | | |
| Respiratory | | | |
| Intra-abdominal | | | |
| Urinary | | | |
| Skin and soft tissue | | | |
| Blood | | | |
| Other | | | |
| Unknown Source | | | |
| Comorbidities | | | |
| 0 | | | |
| 1-2 | | | |
| 3+ | | | |

## Section 6: Analysis

Outcome definitions: List and describe each primary and secondary outcome including details of:

26a specification of outcomes and timings. If applicable include the order of importance of primary or key secondary end points (eg, order in which they will be tested):

Primary outcome: The primary outcome is the proportion of patients achieving either SBP >100 mmHg or MAP > 65 mmHg or a target blood pressure set by the treating physician at 90 (±15) minutes after inclusion.

Secondary outcome A: Number of ICU free days alive within 30 days

Secondary outcome B: Time without shock within 24 hours

Secondary outcome C: 30-day all-cause mortality.

Secondary outcome D: In-hospital all-cause mortality

Tertiary outcome A: Proportion of patients receiving vasopressor at any point within 24 hours.

Tertiary outcome B: Time to vasopressor initiation during hospitalization

Tertiary outcome C: Hours of vasopressor infusion during hospitalization

Tertiary outcome D: Re-admission for any reason within 30 days of inclusion

Tertiary outcome E: ED length of stay

Tertiary outcome F: Proportion of patients admitted to the ICU during hospitalization

Tertiary outcome G: ICU length of stay

Tertiary outcome H: Hospital length of stay

Tertiary outcome I: Need for mechanical ventilation (either invasive or non-invasive ventilation) within 30-days

Tertiary outcome J: Need for renal replacement therapy (continuous renal replacement therapy or dialysis) within 30-days

Tertiary Outcome K: Organ support-free days within 30 days (defined as mechanical ventilation, vasopressor or inotropic therapy, or dialysis)

Tertiary outcome L: Amount of fluid therapy received within the first 24 hours

Safety outcome A: Proportion of patients developing pulmonary oedema within 72 hours (Diagnosed by physician in accordance with local guidelines, e.g., clinical decision including evaluation with paraclinical imaging such as x-ray or lung ultrasound).

Safety outcome B: Proportion of patients developing acute kidney injury within 72 hours (Defined as an absolute increase of creatinine  $\geq 26.5 \mu \text{mol/L}$  or  $\geq 1.5$  fold from baseline)

Safety outcome C: Proportion of patients experiencing extravasation of peripheral noradrenaline

Safety outcome D: Proportion of patients having serious complications due to extravasation (Defined as a serious complication fulfilling the criteria for a serious adverse reaction, e.g. skin necrosis necessitating surgical intervention)

Safety outcome E: Proportion of patients experiencing overdosing due to noradrenaline infusion in the trial (Defined as severe hypertension, and reflex bradycardia suspected by the staff or investigators)

Safety outcome F: Proportion of patients experiencing any SAE, SAR or SUSAR related to the trial intervention or procedures registered during the trial

## 26b specific measurement and units (eg, glucose control, hbA1c [mmol/mol or %])

Measurement units are specified in the protocol available through CTIS under registration 2023-504584-16-00 and codebook (Appendix).

## 26c any calculation or transformation used to derive the outcome (eg, change from baseline, QoL score, time to event, logarithm, etc)

Outcomes that will assess time periods will need to be calculated. This includes, but not limited to, time without shock within 24-hours and number of ICU free days alive within 30 days.

MAP calculations will be performed in the event of missing from the dataset. MAP is not registered as standard if blood pressure targets are entered in the electronic health record. This includes calculation of MAP at ED arrival/triage, which will always be missing. If MAP is present from direct data capture in the trial, this MAP takes precedence and MAP will not be calculated for that registration. All MAP values will be calculated according to the description in section 28: Missing data.

#### Analysis methods

## 27a what analysis method will be used and how the treatment effects will be presented

Primary outcome: The primary outcome is the proportion of patients achieving either SBP >100 mmHg or MAP > 65 mmHg or a target blood pressure set by the treating physician at 90 (±15) minutes after inclusion.

The outcome will be reported as proportions with 95% confidence intervals (CIs) for both arms, and compared by estimating a relative risk (RR) with 95% CIs and p-value by logistic regression followed by prediction of risk via G-computation.

RR and associated 95%CI will be estimated using non-parametric bootstrapping.

Secondary outcome A: Number of ICU free days alive within 30 days

The outcome will be reported as means and mean difference between groups with 95% confidence intervals and compared by linear regression. To take into account the expected non-normality of data, confidence intervals and p-values will be determined by non-parametric bootstrapping.

Secondary outcome B: Time without shock within 24 hours

Secondary outcome C: 30-day all-cause mortality.

Secondary outcome D: In-hospital all-cause mortality

These outcome will be reported as proportions with 95% confidence intervals (CIs) for both arms, and compared by estimating a relative risk (RR) with 95% CIs and p-value by logistic regression followed by prediction of risk via G-computation.

RR and associated 95%CI will be estimated using non-parametric bootstrapping.

Tertiary outcome A: Proportion of patients receiving vasopressor at any point within 24 hours.

Tertiary outcome D: Re-admission for any reason within 30 days of inclusion

Tertiary outcome F: Proportion of patients admitted to the ICU during hospitalization

Tertiary outcome I: Need for mechanical ventilation (either invasive or non-invasive ventilation) within 30-days

Tertiary outcome J: Need for renal replacement therapy (continuous renal replacement therapy or dialysis) within 30-days

These outcome will be reported as proportions with 95% confidence intervals (CIs) for both arms, and compared by estimating a relative risk (RR) with 95% CIs and p-value by logistic regression followed by prediction of risk via G-computation.

RR and associated 95%CI will be estimated using non-parametric bootstrapping.

Tertiary outcome B: Time to vasopressor initiation during hospitalization

Tertiary outcome C: Hours of vasopressor infusion during hospitalization

Tertiary outcome F: Lactate level at study entry

Tertiary outcome I: ED length of stay

Tertiary outcome G: ICU length of stay

Tertiary outcome H: Hospital length of stay

Tertiary Outcome K: Organ support-free days within 30 days (defined as mechanical ventilation, vasopressor or inotropic therapy, or dialysis)

Tertiary outcome L: Amount of fluid therapy received within the first 24 hours

These outcomes will be reported as means and mean difference between groups with 95% confidence intervals and compared by linear regression. To take into account the expected non-normality of data, confidence intervals and p-values will be determined by non-parametric bootstrapping.

Safety outcome A: Proportion of patients developing pulmonary oedema within 72 hours (Diagnosed by physician in accordance with local guidelines, e.g., clinical decision including evaluation with paraclinical imaging such as x-ray or lung ultrasound).

Safety outcome B: Proportion of patients developing acute kidney injury within 72 hours (Defined as an absolute increase of creatinine  $\geq$ 26.5 $\mu$ mol/L or  $\geq$ 1.5 fold from baseline)

Safety outcome C: Proportion of patients experiencing extravasation of peripheral noradrenaline

Safety outcome D: Proportion of patients having serious complications due to extravasation (Defined as a serious complication fulfilling the criteria for a serious adverse reaction, e.g. skin necrosis necessitating surgical intervention)

Safety outcome E: Proportion of patients experiencing overdosing due to noradrenaline infusion in the trial (Defined as severe hypertension, and reflex bradycardia suspected by the staff or investigators)

Safety outcome F: Proportion of patients experiencing any SAE, SAR or SUSAR related to the trial intervention or procedures registered during the trial

These outcomes will be reported as proportions with 95% confidence intervals (CIs) for both arms, and compared by estimating a relative risk (RR) with 95% CIs and p-value by logistic regression followed by prediction of risk via G-computation.

RR and associated 95%CI will be estimated using non-parametric bootstrapping.

#### 27b any adjustment for covariates

All parameters in the main analysis will be adjusted for baseline covariates of age (divided in age groups of 18-29, 30-39, 40-49, 50-59, 60-69, 70-79, 80-89, 90+), lactate at inclusion (<2,  $\ge 2$  - <4,  $\ge 4$ ) and trial site.

#### 27c methods used for assumptions to be checked for statistical methods

Distributional assumptions on bootstraps and G-computation will be investigated by quantile-quantile plots.

27d details of alternative methods to be used if distributional assumptions do not hold, eg, normality, proportional hazards, etc

If bootstrapping of linear regression deviates markedly from distributional assumption, a quantile regression estimating the median, and median differences instead of mean and mean differences will be performed.

## 27e any planned sensitivity analyses for each outcome where applicable

All outcomes will be reanalyzed as a per-protocol analysis.

Due to the nature of the pragmatic trial design, only participants in the intervention group not receiving vasopressors in the ED are expected to influence the analysis groups in the per-protocol analysis. All standard care groups are expected to receive standard care.

#### 27f any planned subgroup analyses for each outcome including how subgroups are defined

The substudies will be analysed including only those participants included in each substudy. Details on substudies are not part of this SAP.

No additional subgroup analyses are planned.

## Missing data

#### 28 Reporting and assumptions/statistical methods to handle missing data (e.g., multiple imputation)

Missing data will be reported in all relevant publications. We do not expect missing data regarding the primary outcome of the trial or key secondary outcomes. We do expect some missing data in the variables for calculating some outcomes, including the secondary outcomes, as well as missing data or loss to follow-up for the long-term outcomes in the trial. We do not expect missing data for AE or SAE.

No imputation or weighting of missing data is planned, as only a small number of missing data is expected with the following exception:

MAP values are not always registered as part of the electronic health records, as the standard is to register systolic and diastolic blood pressure, unless patients are monitored in the intensive care unit. This provides a potential substantial number of missing MAP values, especially for patients who are not receiving the intervention in the intervention group at the time of measurement, or patients who are not admitted to the ICU. For non-invasive measurements, the measured MAP values can be imprecise, especially in the event of hypotension, due to how the measurement method obtains the blood pressure values. It can therefore overestimate parameters.

We will perform imputation of missing MAP values, if the MAP is missing but systolic (SBP) and diastolic blood pressure (DBP) are present, for all timepoints during the trial. Imputation will be performed using predictive mean matching. A maximum value of each blood pressure measurement at each specific timepoint will initially be calculated using the standard formula for calculating MAP using Systolic (SBP) and Diastolic Blood Pressure (DBP):

$$MAP = \frac{2 * DBP + SBP}{3}$$

If the imputed measurement is above this calculated MAP, the calculated MAP will be used. If it is below the calculated MAP value, the imputed measurement will be used.

This data imputation is only expected to be relevant for calculating the key secondary outcome of time without shock within 24 hours. It will not apply to the primary outcome.

#### Additional analyses

## 29 Details of any additional statistical analyses required, eg, complier-average causal effect analysis

We will perform a Bayesian sensitivity analysis of the primary and secondary outcomes, following the same methodology as the main analyses. Based on this analysis we will report posterior probabilities for a range of effect sizes. The Bayesian analyses will utilize weakly informative priors, symmetric with respect to the intervention.

#### Harms

30 Sufficient details on summarizing safety data, e.g., information on severity, expectedness, and causality; details of how adverse events are coded or categorized; how adverse event data will be analysed, i.e., grade 3/4 only, incidence case analysis, intervention emergent analysis

Harms are presented partly as tertiary/explorative outcomes as presented in Section 6: Analysis.

Details on harms and safety are available in section 7 in the protocol.

#### Statistical software

#### 31 Details of statistical packages to be used to carry out analyses

Statistical analyses will be performed using R 4.4.5 (R Core Team 2024, Vienna) or a newer version, if such is published before the analyses. The version used will be reported in the manuscript.

## References

## 32a References to be provided for nonstandard statistical methods

G-computation: Naimi AI, Cole SR, Kennedy EH. An introduction to g methods. Int J Epidemiol. 2017;46(2):756-62.Bayesian Analysis: Gelman A, Carlin JB, Stern HS, Dunson DB, Vehtari A, Rubin DB. Bayesian Data Analysis. 3rd ed2013.

#### 32b Reference to Data Management Plan

See section 9 in the protocol.

The codebook for the REDCap database which includes definition and validation of variables collected in the trial are available as a supplementary file.

#### 32c Reference to the Trial Master File and Statistical Master File

The Trial Master File exist partly as a physical folder in the Emergency Department at Odense University Hospital and partly as an electronic version located in a secure SharePoint server under The Region of Southern Denmark. The Trial Master File can be accessed with appropriate and necessary agreement with the Sponsor.

#### 32d Reference to other standard operating procedures or documents to be adhered to

Gamble C, Krishan A, Stocken D, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA 2017;318(23):2337-2343. DOI: 10.1001/jama.2017.18556

#### 32e References to other litterature

- 1. Gamble C, Krishan A, Stocken D, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA 2017;318(23):2337-2343. DOI: 10.1001/jama.2017.18556.
- 2. Gitz Holler J, Jensen HK, Henriksen DP, et al. Etiology of Shock in the Emergency Department: A 12-Year Population-Based Cohort Study. Shock 2019;51(1):60-67. DOI: 10.1097/SHK.00000000000816.
- 3. Vincent JL, De Backer D. Circulatory shock. N Engl J Med 2013;369(18):1726-34. DOI: 10.1056/NEJMra1208943.
- 4. Holler JG, Bech CN, Henriksen DP, Mikkelsen S, Pedersen C, Lassen AT. Nontraumatic hypotension and shock in the emergency department and the prehospital setting, prevalence, etiology, and mortality: a systematic review. PLoS One 2015;10(3):e0119331. DOI: 10.1371/journal.pone.0119331.
- 5. Finfer S, Liu B, Taylor C, et al. Resuscitation fluid use in critically ill adults: an international cross-sectional study in 391 intensive care units. Crit Care 2010;14(5):R185. DOI: 10.1186/cc9293.
- 6. Jessen MK, Simonsen BY, Thomsen MH, Andersen LW, Kolsen-Petersen JA, Kirkegaard H. Fluid management of emergency department patients with sepsis-A survey of fluid resuscitation practices. Acta Anaesthesiol Scand 2022;66(10):1237-1246. DOI: 10.1111/aas.14141.
- 7. Jessen MK, Andersen LW, Thomsen MH, et al. Twenty-four-hour fluid administration in emergency department patients with suspected infection: A multicenter, prospective, observational study. Acta Anaesthesiol Scand 2021;65(8):1122-1142. DOI: 10.1111/aas.13848.
- 8. Marik PE, Linde-Zwirble WT, Bittner EA, Sahatjian J, Hansell D. Fluid administration in severe sepsis and septic shock, patterns and outcomes: an analysis of a large national database. Intensive Care Med 2017;43(5):625-632. DOI: 10.1007/s00134-016-4675-y.
- 9. National Heart L, Blood Institute Acute Respiratory Distress Syndrome Clinical Trials N, Wiedemann HP, et al. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med 2006;354(24):2564-75. DOI: 10.1056/NEJMoa062200.
- 10. Silversides JA, Major E, Ferguson AJ, et al. Conservative fluid management or deresuscitation for patients with sepsis or acute respiratory distress syndrome following the resuscitation phase of critical illness: a systematic review and meta-analysis. Intensive Care Medicine: Springer Verlag; 2017:155-170.
- 11. Perner A, Cecconi M, Cronhjort M, et al. Expert statement for the management of hypovolemia in sepsis. Intensive Care Medicine: Springer Verlag; 2018:791-798.
- 12. National Heart L, Blood Institute P, Early Treatment of Acute Lung Injury Clinical Trials N, et al. Early Restrictive or Liberal Fluid Management for Sepsis-Induced Hypotension. N Engl J Med 2023;388(6):499-510. DOI: 10.1056/NEJMoa2212663.
- 13. Evans L, Rhodes A, Alhazzani W, et al. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 20212021.

- 14. Djogovic D, Macdonald S, Wensel A, et al. Vasopressor and inotrope use in canadian emergency departments: Evidence based consensus guidelines. Canadian Journal of Emergency Medicine: Decker Publishing; 2015:1-16.
- 15. Self WH, Semler MW, Bellomo R, et al. Liberal Versus Restrictive Intravenous Fluid Therapy for Early Septic Shock: Rationale for a Randomized Trial. Ann Emerg Med 2018;72(4):457-466. DOI: 10.1016/j.annemergmed.2018.03.039.
- 16. Ospina-Tascón GA, Hernandez G, Bakker J. Should we start vasopressors very early in septic shock? Journal of Thoracic Disease 2020;12(7):3893-3896. DOI: 10.21037/jtd.2020.02.21.
- 17. Russell JA. Vasopressor therapy in critically ill patients with shock. Intensive Care Med 2019;45(11):1503-1517. DOI: 10.1007/s00134-019-05801-z.
- 18. Tian DH, Smyth C, Keijzers G, et al. Safety of peripheral administration of vasopressor medications: A systematic review. Emerg Med Australas 2020;32(2):220-227. DOI: 10.1111/1742-6723.13406.
- 19. Black LP, Puskarich MA, Smotherman C, Miller T, Fernandez R, Guirgis FW. Time to vasopressor initiation and organ failure progression in early septic shock. J Am Coll Emerg Physicians Open 2020;1(3):222-230. DOI: 10.1002/emp2.12060.
- 20. Colon Hidalgo D, Patel J, Masic D, Park D, Rech MA. Delayed vasopressor initiation is associated with increased mortality in patients with septic shock. J Crit Care 2020;55:145-148. DOI: 10.1016/j.jcrc.2019.11.004.
- 21. Delaney A, Finnis M, Bellomo R, et al. Initiation of vasopressor infusions via peripheral versus central access in patients with early septic shock: A retrospective cohort study. Emerg Med Australas 2020;32(2):210-219. DOI: 10.1111/1742-6723.13394.
- 22. Keijzers G, Macdonald SP, Udy AA, et al. The Australasian Resuscitation In Sepsis Evaluation: Fluids or vasopressors in emergency department sepsis (ARISE FLUIDS), a multi-centre observational study describing current practice in Australia and New Zealand. Emerg Med Australas 2020;32(4):586-598. DOI: 10.1111/1742-6723.13469.
- 23. Tank AW, Lee Wong D. Peripheral and central effects of circulating catecholamines. Compr Physiol 2015;5(1):1-15. DOI: 10.1002/cphy.c140007.
- 24. Permpikul C, Tongyoo S, Viarasilpa T, Trainarongsakul T, Chakorn T, Udompanturak S. Early Use of Norepinephrine in Septic Shock Resuscitation (CENSER). A Randomized Trial. Am J Respir Crit Care Med 2019;199(9):1097-1105. DOI: 10.1164/rccm.201806-1034OC.
- 25. Araiza A, Duran M, Varon J. Administration of vasopressors through peripheral venous catheters. CMAJ 2022;194(21):E739. DOI: 10.1503/cmaj.211966.
- 26. Gamper G, Havel C, Arrich J, et al. Vasopressors for hypotensive shock. Cochrane Database of Systematic Reviews: John Wiley and Sons Ltd; 2016.
- 27. Lewis T, Merchan C, Altshuler D, Papadopoulos J. Safety of the Peripheral Administration of Vasopressor Agents. J Intensive Care Med 2019;34(1):26-33. DOI: 10.1177/0885066616686035.
- 28. Loubani OM, Green RS. A systematic review of extravasation and local tissue injury from administration of vasopressors through peripheral intravenous catheters and central venous catheters. J Crit Care 2015;30(3):653 e9-17. DOI: 10.1016/j.jcrc.2015.01.014.

- 29. Tran QK, Mester G, Bzhilyanskaya V, et al. Complication of vasopressor infusion through peripheral venous catheter: A systematic review and meta-analysis. American Journal of Emergency Medicine: W.B. Saunders; 2020.
- 30. Lewis SR, Pritchard MW, Evans DJ, et al. Colloids versus crystalloids for fluid resuscitation in critically ill people. Cochrane Database Syst Rev 2018;8(8):CD000567. DOI: 10.1002/14651858.CD000567.pub7.
- 31. Nguyen TT, Surrey A, Barmaan B, et al. Utilization and extravasation of peripheral norepinephrine in the emergency department. Am J Emerg Med 2021;39:55-59. DOI: 10.1016/j.ajem.2020.01.014.
- 32. Gamerman V, Cai T, Elsäßer A. Pragmatic randomized clinical trials: best practices and statistical guidance. Health Services and Outcomes Research Methodology 2019;19(1):23-35. DOI: 10.1007/s10742-018-0192-5.
- 33. Zwarenstein M, Treweek S, Gagnier JJ, et al. Improving the reporting of pragmatic trials: An extension of the CONSORT statement. Bmj 2008;337(7680):1223-1226. DOI: 10.1136/bmj.a2390.
- 34. Harris PA, Taylor R, Minor BL, et al. The REDCap consortium: Building an international community of software platform partners. Journal of Biomedical Informatics 2019;95(April):103208-103208. DOI: 10.1016/j.jbi.2019.103208.
- 35. Schulz KF, Altman DG, Moher D, Group C. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ 2010;340(7748):c332. DOI: 10.1136/bmj.c332.

## **Appendix**

## Appendix 1: CONSORT diagram draft

